CLINICAL TRIAL: NCT07276633
Title: Effect of Subanesthetic Dose Propofol Use Before Extubation on Recovery From Anesthesia, Agitation on Recovery, and Patient Satisfaction
Brief Title: Use of Subanesthetic Dose Propofol Before Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Associate professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Subanesthetic Dose of Propofol
Record Dates: First submitted 2025-11-16; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2024-05

CONDITIONS: Emergence Agitation; Rhinoplasty; Patient Satisfaction
Keywords: Propofol; Postoperative Recovery; Patient Satisfaction; Emergence Agitation; Rhinoplasty; General Anesthesia Recovery; Sub-Anesthetic Dose
MeSH Terms: conditions — Emergence Delirium; Patient Satisfaction | interventions — Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol Group (Active Comparator): Sub-anesthetic dose of propofol (0.5 mg/kg) administered 10 minutes before extubation.
  Interventions: Other: Normal Saline (Placebo)
- Control Group (Sham Comparator): Normal saline administered 10 minutes before extubation.
  Interventions: Drug: Propofol (Sub-Anesthetic Dose)

INTERVENTIONS:
Drug: Propofol (Sub-Anesthetic Dose) — Participants receive 0.5 mg/kg intravenous propofol as a single bolus 10 minutes before extubation.
  Other Names: Normal saline administered pre-extubation
  Arms: Control Group
Other: Normal Saline (Placebo) — Participants receive an equivalent volume of normal saline 10 minutes before extubation.
  Arms: Propofol Group

SUMMARY:
This study investigates whether administering a low, sub-anesthetic dose of propofol before extubation can reduce emergence agitation and improve perioperative comfort in patients undergoing rhinoplasty. Emergence agitation refers to restlessness and confusion during early recovery from anesthesia, which may affect patient safety and surgical conditions. The study evaluates agitation levels, recovery characteristics, and patient-reported comfort following propofol administration compared with standard care.

DETAILED DESCRIPTION:
This study aims to evaluate whether administering a sub-anesthetic dose of propofol before extubation can reduce emergence agitation, enhance recovery characteristics, and improve patient comfort in adults undergoing rhinoplasty surgery. Emergence agitation is a common phenomenon during early recovery from general anesthesia and can involve restlessness, disorientation, and involuntary movements, potentially affecting patient safety and surgical outcomes. The study uses a randomized controlled design to compare peri-extubation responses between patients receiving low-dose propofol and those receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* Patients scheduled for rhinoplasty surgery
* ASA physical status I-II
* No respiratory tract infection
* Provided written informed consent

Exclusion Criteria:

* Refusal to participate
* Presence of any respiratory tract infection
* Younger than 18 or older than 65
* ASA III-IV
* Known allergy to study medications
* Predicted difficult intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Changing Preoperative Anxiety Score (STAI) | 15 minutes (T1-T2)
  Comparison of the State-Trait Anxiety Inventory (STAI) state anxiety score measured in the preoperative waiting room (T1) with the STAI score 15 minutes after the palming technique (T2). The difference between the two time points is analyzed to assess the anxiety-reducing effect of the intervention.

SECONDARY OUTCOMES:
Hemodynamic Parameter Changes | 15 minutes (T1-T2)
  Changes in heart rate (HR) values between the T1 and T2 time points. The effect of the palming technique on hemodynamic stability is evaluated.
Hemodynamic Parameter Changes | 15 minutes (T1-T2)
  Changes in mean blood pressure values between the T1 and T2 time points. The effect of the palming technique on hemodynamic stability is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yuzkat, Associate professor, Principal Investigator — Yuzuncu Yil University Dursun Odabas Medical Center
Locations (1):
- Yuzuncu Yil University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available because data sharing was not included in the informed consent and sharing such data could compromise patient confidentiality.

REFERENCES:
- [Background] Kanaya A, Kuratani N, Satoh D, Kurosawa S. Lower incidence of emergence agitation in children after propofol anesthesia compared with sevoflurane: a meta-analysis of randomized controlled trials. J Anesth. 2014 Feb;28(1):4-11. doi: 10.1007/s00540-013-1656-y. Epub 2013 Jun 26. PMID 23800983